CLINICAL TRIAL: NCT02914548
Title: A Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Comparison Trial to Assess the Efficacy and Safety of 0.3% and 1% OPA-15406 Ointments in Patients With Atopic Dermatitis
Brief Title: Study of OPA-15406 Ointment in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 271-15-001; JapicCTI-163372 (Other: Japic)
Record Dates: First submitted 2016-09-08; First posted 2016-09-26 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.3% OPA-15406 (Experimental): Subjects were treated with assigned 0.3% OPA-15406 ointment twice daily.
  Interventions: Drug: OPA-15406
- 1% OPA-15406 (Experimental): Subjects were treated with assigned 1% OPA-15406 ointment twice daily.
  Interventions: Drug: OPA-15406
- Placebo (Placebo Comparator): Subjects were treated with assigned 0% OPA-15406 ointment twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPA-15406 — Subjects were treated with assigned 0.3% or 1% OPA-15406 ointment twice daily.
  Arms: 0.3% OPA-15406; 1% OPA-15406
Drug: Placebo — Subjects were treated with assigned 0% OPA-15406 ointment twice daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of OPA-15406 ointment in patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atopic dermatitis based on the criteria of Hanifin and Rajka

Exclusion Criteria:

* Subjects who have an atopic dermatitis or contact dermatitis flare-up defined as a sudden intensification of atopic dermatitis.
* Subjects who have an active viral skin infection.
* Subjects with a current or history of malignancy.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (3):
- Japan (3):
  - Hokkaido Region
  - Kanto Region
  - Kiniki Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
Started | 67 | 67 | 66
Completed | 46 | 53 | 46
Not Completed | 21 | 14 | 20
Not completed — Adverse Event | 15 | 7 | 15
Not completed — Physician Decision | 2 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 4
Not completed — >40% of body surface area | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo | Total
Number analyzed (Participants) | 67 | 67 | 66 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 1 | 3
  Between 18 and 65 years | 65 | 67 | 65 | 197
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (9.0) | 31.0 (10.8) | 31.6 (10.0) | 30.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 23 | 70
  Male | 45 | 42 | 43 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 67 | 67 | 66 | 200
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 67 | 67 | 66 | 200

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate of Investigator's Global Assessment(IGA) of Disease Severity at Week4
Description: The investigator or sub investigator assessed the skin symptoms using IGA. The investigator or sub investigator scored the severity (0 = clear, 1 = almost clear, 2 =mild, 3 = moderate, 4 = severe/very severe) of the overall symptoms of the treatment area (erythema, infiltration, papules, effusion and scab formation) from baseline to Week4. Incidence of success in IGA was defined as the rate of subjects whose IGA score was 0 (clear) or 1 (almost clear) and had improved by at least 2 grades (responders) from baseline.
Time Frame: At Week 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 67 | 67 | 66
percentage of participants | 14.93 [7.40 to 25.74] | 22.39 [13.11 to 34.22] | 9.09 [3.41 to 18.74]

2. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: The investigator or sub investigator assessed the symptoms of AD using EASI. EASI's minimum and maximum scores are 0 and 72 scores respectively. The higher the EASI score is, the more severe the symptoms of AD, and a negative change from the baseline means improvement and a positive change means worsening. The investigator or sub investigator scored the severity (0-3 points) and affected BSA (%) based on the 4 symptoms (erythema, infiltration/papules, excoriation, and lichenification) on the 4 body regions (face, neck and head ; upper limbs ;trunk; and lower limbs). Number of participants analyzed represents number of participants with data at both Baseline and Week4. Participants who have no data were excluded.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 57 | 58 | 53
score on a scale | -2.32 (0.75) | -3.16 (0.75) | -0.15 (0.77)

3. Secondary Outcome: Change From Baseline in Visual Analogue Scale(VAS) for Pruritus Score
Description: The investigator or subinvestigator evaluated the level of pruritus based on VAS. The subjects will mark the point of pruritus intensity during the last 24 hours on the line of a 100- mm VAS sheet between the left end (no pruritus: the score is 0 ) and the right end (very severe pruritus: the score is 100), and a negative change from the baseline means improvement and a positive change means worsening. Number of participants analyzed represents number of participants with data at both Baseline and Week4. Participants who have no data were excluded
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: mm
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 57 | 58 | 53
mm | -6.76 (3.31) | -6.28 (3.32) | 0.90 (3.24)

4. Secondary Outcome: Change From Baseline in Verbal Rating Scale(VRS) for Pruritus Score
Description: The investigator or subinvestigator evaluated the pruritus intensity based on VRS. The subjects aged 7 to 14 years old evaluated the pruritus intensity according to the following criteria. The subjects recorded the level of pruritus and the time and date of evaluation in a pruritus diary.
  0 : None
  1. : Mild
  2. : Moderate
  3. : Severe For subjects aged 2 to 6 years, this would not be evaluated. Number of participants analyzed represents number of participants with data at both Baseline and Week4. Participants who have no data were excluded.
Time Frame: Baseline, Hour 156
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 55 | 54 | 47
score on a scale | -0.43 (0.10) | -0.49 (0.10) | -0.06 (0.10)

5. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure(POEM) Score
Description: The investigator or sub investigator evaluated eczema according to the POEM. The subjects answered 7 questions about their eczema by 0-4 points per question. The POEMS's minimum and maximum scores are 0 and 28 scores respectively. The higher the POEM score is, the more severe the symptoms are, and a negative change from the baseline means improvement and a positive change means worsening. If it is difficult for subjects to answer the questions, their parents answered them instead. Number of participants analyzed represents number of participants with data at both Baseline and Week4. Participants who have no data were excluded.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 57 | 58 | 53
score on a scale | -1.36 (0.77) | -2.90 (0.76) | -0.02 (0.79)

6. Secondary Outcome: Change From Baseline in Percentage Affected Body Surface Area
Description: The investigator or subinvestigator drew the affected BSA (range of skin eruption at the time of examination) on the human body drawing to determine the affected areas (%) on the respective 4 body regions (face, neck, and head; upper limbs; trunk; and lower limbs). One palm of the subject corresponds to 1% BSA.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: percentage of Affected Body Surface Area
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
Number analyzed (Participants) | 57 | 58 | 53
percentage of Affected Body Surface Area | -3.94 (1.44) | -3.73 (1.43) | -0.32 (1.48)

7. Secondary Outcome: Mean (SD) OPA-15406 Plasma Trough Concentrations
Description: The plasma concentration of OPA-15406 was measured at Week1, Week4 and Week8. On the day of measurement, the subjects visited the trial site without morning Investigational Medicinal Product (IMP) administration.
  Number of participants analyzed represents number of participants with data at each point. Participants who have no effective data were excluded.
Time Frame: Week1, Week4, Week8
Population: All subjects who had received the IMP at least once and whose plasma drug concentration had been measured
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 64 | 62
ng/mL/mg
  Week 1: number analyzed (Participants) | 53 | 59
  Week 1 | 1.74 (1.87) | 4.96 (5.04)
  Week 4: number analyzed (Participants) | 49 | 50
  Week 4 | 1.71 (2.50) | 5.22 (4.70)
  Week 8: number analyzed (Participants) | 43 | 46
  Week 8 | 1.51 (1.77) | 5.52 (8.28)

8. Secondary Outcome: Mean (SD) Normalized OPA-15406 Plasma Trough Concentrations by Dose Derived From %BSA
Description: The plasma concentration of OPA-15406 was measured at Week1, Week4 and Week8. On the day of measurement, the subjects visited the trial site without morning Investigational Medicinal Product (IMP) administration.Number of participants analyzed represents number of participants with data at each point. Participants who have no effective data were excluded.
Time Frame: Week1, Week4, Week8
Population: All subjects who had received the IMP at least once and whose plasma drug concentration had been measured
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 64 | 62
ng/mL/mg
  Week 1: number analyzed (Participants) | 53 | 59
  Week 1 | 0.114 (0.0991) | 0.113 (0.0952)
  Week 4: number analyzed (Participants) | 49 | 50
  Week 4 | 0.104 (0.119) | 0.127 (0.119)
  Week 8: number analyzed (Participants) | 43 | 46
  Week 8 | 0.0910 (0.103) | 0.137 (0.242)

9. Secondary Outcome: OPA-15406 Plasma PK Parameters, Cmax
Description: OPA-15406 plasma PK parameter (Cmax) was measured on Day 1 and at Week 4 following topical administration of OPA-15406 0.3% and 1% ointment to adult subjects with AD.Number of participants analyzed represents number of participants with effective data at each point. Participants who have no effective data were excluded.
Time Frame: Day 1 and Week 4
Population: All subjects who had received the IMP at least once and whose plasma drug concentration had been measured
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 11 | 9
ng/mL
  Day 1 | 4.01 (5.90) | 7.27 (6.42)
  Week 4: number analyzed (Participants) | 8 | 6
  Week 4 | 2.07 (1.47) | 10.4 (3.68)

10. Secondary Outcome: OPA-15406 Plasma PK Parameters, AUC8h
Description: OPA-15406 plasma PK parameter (AUC8h) was measured on Day 1 and at Week 4 following topical administration of OPA-15406 0.3% and 1% ointment to adult subjects with AD.Number of participants analyzed represents number of participants with effective data at each point. Participants who have no effective data were excluded.
Time Frame: Day 1 and Week 4
Population: All subjects who had received the IMP at least once and whose plasma drug concentration had been measured
Measure: Mean (Standard Deviation); unit: ng・h/mL
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 11 | 9
ng・h/mL
  Day 1 | 22.0 (34.7) | 41.6 (37.6)
  Week 4: number analyzed (Participants) | 8 | 6
  Week 4 | 11.6 (7.23) | 65.2 (26.8)

ADVERSE EVENTS:
Time Frame: Treatment period (8 weeks)
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/66
Other Adverse Events (participants affected / at risk) | 22/67 | 11/67 | 20/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% OPA-15406 (N=67) | 1% OPA-15406 (N=67) | Placebo (N=66)
Viral upper respiratory tract infection (Infections and infestations) | 7 | 4 | 7
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 | 6 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT02914548/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02914548/SAP_001.pdf